CLINICAL TRIAL: NCT04719299
Title: Effectiveness of Smartphone Application in Reducing Anxiety During Pediatric Dental Procedures: a Controlled Clinical Study
Brief Title: Smartphone Application in Reducing Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TPD
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smart phone application (Experimental): Behavior modification of patients will be done by showing them smartphone application game. The game demonstrates the use of common dental equipment like mirrors, ultrasonic scalers, handpieces and suction tips, etc. in the form of animated pictures with visual and sound effects. The dentist will play the game to show the child the dental procedure that will be performed on him later.
  Interventions: Behavioral: Tell-Play-Do
- traditional behavior management technique (Active Comparator): Using traditional behavior management techniques (Tell-Show-Do) which will be applied prior to local anesthesia administration
  Interventions: Behavioral: Tell-Show-Do

INTERVENTIONS:
Behavioral: Tell-Play-Do — Using smart phone application
  Arms: smart phone application
Behavioral: Tell-Show-Do — Using traditional behavior management technique
  Arms: traditional behavior management technique

SUMMARY:
evaluating the effectiveness of smartphone applications (Tell-Play-Do) (TPD) in reduction of preoperative anxiety in children undergoing restorative treatment, as measured by heart rate and Venham's Picture Test.

DETAILED DESCRIPTION:
A total of at least 78 patients aged from 6-8 years will be included. All participants will be divided equally into two groups. Study group TPD using smartphone application and Control group (Tell-Show-Do) (TSD) using traditional behavior management technique.

Dental anxiety using Venham's Picture Test and heart rate using pulse oximeter will be assessed during dental treatment

ELIGIBILITY:
Inclusion Criteria:

* School-age children aged from 6-8 years.
* Presence of carious primary molars without pulpal involvement.
* Parents have the ability to write, read and willingness to participate in the study.
* First dental visit to the clinic.
* Normal healthy children.

Exclusion Criteria:

* Children with previous dental experience.
* Medically compromised children.
* Children with special needs (physical or mental).

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2020-12-27 (Actual)

PRIMARY OUTCOMES:
Change in dental anxiety scores | Baseline and immediate post operative
  The number of times the "anxious" figure will be chosen a score of one will be assigned and then totaled to give a final score (minimum score - zero; maximum score - eight) for each patient.
  The final score will be interpreted as follow: 8 (Very high anxiety), Equal to or more than 6 and less than 8 (High anxiety), Equal to or more than 4 and less than 6 (Average), Equal to or more than 2 and less than 4 (Low anxiety), More than 0 and less than 2 (Very low anxiety) and 0 (No anxiety).
Change in heart rate | Baseline and immediate post operative
  recorded by using pulse oximeter as a potential secondary measure of anxiety (physiological parameter).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt